CLINICAL TRIAL: NCT01314599
Title: Open-Label, Dose-Escalating, Clinical and Pharmacokinetic Phase I Study of Lurbinectedin (PM01183) in Patients With Advanced Acute Leukemia or Relapsed/Refractory Myelodysplastic Syndrome.
Brief Title: Clinical Study of PM01183 in Patients With Acute Leukemia or Relapsed/Refractory Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PM1183-A-002-10
Record Dates: First submitted 2011-03-09; First posted 2011-03-14 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-07

CONDITIONS: Acute Leukemia
Keywords: Leukemia; lurbinectedin; PM01183; Pharma Mar; Acute Leukemia in Relapse and Primary Refractory
MeSH Terms: conditions — Leukemia | interventions — PM 01183; Powders; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): PM01183 will be administered i.v. as a 1-hour infusion through a pump device at escalating doses according to the respective dose level, on Days 1 and 8 of each treatment phase.
  Interventions: Drug: PM01183 1 mg Powder for concentrate for solution for infusion and PM01183 4 mg Powder for concentrate for solution for infusion

INTERVENTIONS:
Drug: PM01183 1 mg Powder for concentrate for solution for infusion and PM01183 4 mg Powder for concentrate for solution for infusion — PM01183 Drug Product will be provided as a lyophilized powder for concentrate for solution for infusion with a strength of 1.0 mg/vial and 4.0 mg/vial.
  Before use, the vials will be reconstituted with 2 ml or 8 ml of sterile water for injection to give a solution containing 0.5 mg/ml of PM01183.

SUMMARY:
Phase I Study of PM01183 in Patients with Advanced Acute Leukemia to determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM01183.

DETAILED DESCRIPTION:
Open-Label, Dose-Escalating, Clinical and Pharmacokinetic Phase I Study of PM01183 in Patients with Advanced Acute Leukemia to determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM01183 administered as 1-hour intravenous (i.v.) infusion on three consecutive days (Days 1-3) to patients with advanced acute leukemia and to assess the safety profile and tolerability, to obtain preliminary information on the efficacy and to characterize the pharmacokinetics (PK) and pharmacogenomic (PGx) profile of PM01183.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed and dated written informed consent
* Age ≥ 18 years.
* Patients must have a previous cytological or histological diagnosis of:

  * Relapsed or primary refractory non-M3 acute myeloid leukemia (AML) by the World Health Organization (WHO) criteria (irrespective of the number of prior regimens), either de novo or secondary [i.e., secondary to myelodysplastic syndromes (MDS), myeloproliferative neoplasms or previous chemotherapy for another condition].
  * Untreated AML in patients ≥ 65 years of age, if patients are not candidates for standard induction chemotherapy or have poor risk AML (i.e., secondary AML or AML with adverse cytogenetics or complex karyotype).
  * Accelerated or blastic phase chronic myeloid leukemia (CML, with progressive disease despite treatment with BCR-ABL kinase inhibitors), or chronic myelomonocytic leukemia (CMML).
  * Relapsed or refractory acute lymphoblastic leukemia (ALL) by WHO criteria.
* Patients must have the following laboratory values prior to the start of treatment:

  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) range of values, unless due to elevated indirect bilirubin (e.g.,Gilbert's syndrome or hemolysis).
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN.
  * Alkaline phosphatase (AP) ≤ 2.5 x ULN.
  * Albumin ≥ 2.5 g/dl.
  * Calculated creatinine clearance (CrCl) ≥ 30 ml/min (using Cockcroft and Gault's formula).
  * Creatine phosphokinase (CPK) ≤ 2.5 x ULN.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

* Pregnant or lactating women; men and women of reproductive potential who are not using effective contraceptive methods throughout the treatment period and for six months after discontinuation of treatment.
* Patients who plan to undergo allogeneic BM transplantation within four weeks.
* Other relevant diseases or adverse clinical conditions:

  * History or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically significant valvular heart disease within last year.
  * Symptomatic or unstable cardiac arrhythmias, and/or prolonged QT-QTc grade ≥ 2.
  * History of significant neurological or psychiatric disorders that may affect the patient's compliance with the protocol assessments.
  * Active uncontrolled infection.
  * Myopathy or any clinical situation that causes significant and persistent elevation of CPK (> 2.5 x ULN in two different determinations performed one week apart).
  * Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis).
  * Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
* Hematopoietic allogeneic stem cell transplantation within the last four months and/or active graft versus host disease, or prior autologous transplantation within the last four weeks.
* Patients known to be human immunodeficiency virus (HIV) positive.
* Cytotoxic chemotherapy within the last two weeks; radiation therapy within the last two weeks; biologic agents, including hematopoietic growth factors, within the last week; hydroxyurea, imatinib, corticosteroids and arsenic trioxide should be discontinued at least 24 hours prior to first study drug administration.
* Treatment with any investigational product in the ≤ 5 half-lives period prior to inclusion in the study, or 30 days after therapy (in case of unknown half-life), unless evidence of rapid proliferating disease and upon discussion with the Sponsor.
* Known hypersensitivity to any of the components of the drug product (DP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Dose (RD) of PM01183 in patients with advanced acute leukemia. | Up to 30 months
  The recommended dose (RD) will be the immediate lower DL below the MTD (maximum tolerated dose)with less than 1/3 of the first 6 evaluable patients experiencing DLT (dose limiting toxicity)during the induction, provided the RD is ≥ dose level 2. If the RD is determined at dose level 1, no further expansion will be done, and the study will be terminated.

SECONDARY OUTCOMES:
Antileukemic activity | After induction/reinduction and every 4 weeks after treatment discontinuation; up to 30 months
  Activity will be defined according to the International Working Group (IWG) criteria.
Pharmacogenomic (PGx) profile of PM01183 in patients with advanced acute leukemia. | Between day -24 to day 1
  Identification of potential biomarkers of response to PM01183
Pharmacokinetics (PK) of PM01183 in patients with advanced acute leukemia | Days 1 to 8 of induction and day 1 of next phase
  The PK will be elucidated using standard non-compartmental methods. The following parameters will be calculated: maximum drug concentration (Cmax), area under the curve (AUC), volume of distribution based on the terminal half-life (Vz), volume of distribution at steady state (Vss), clearance (CL) and half-life (t1/2)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rochester, Minnesota
  - Houston, Texas